CLINICAL TRIAL: NCT05889429
Title: Correlation Between Brain Structure and Activity and Spontaneous Recovery of Motor Function Following Brain Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technion, Israel Institute of Technology (Other)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Firas Mawase, Prof. Firas Mawase, Technion, Israel Institute of Technology
Other Study IDs: MOH_2020-06-24_009069
Record Dates: First submitted 2023-05-09; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- brain ischemic stroke patients: Participants who meet the inclusion criteria.
  All participants will undergo four testing sessions spanning the acute and subacute post-stroke phases:
  Session 1 (t1) - 2-14 days from stroke onset Session 2 (t2) - 4 weeks (± 7 days) after the stroke Session 3 (t3) - 8 weeks (± 7 days) after the stroke Session 4 (t4) - 12 weeks (± 7 days) after the stroke
  Interventions: Diagnostic Test: MRI scans; Behavioral: clinical assessments
- Control group: Participants with healthy age and gender-matched with no history of neurological impairments.
  Each participant will visit the testing sites 4 times within one month between different sessions.
  Interventions: Diagnostic Test: MRI scans

INTERVENTIONS:
Diagnostic Test: MRI scans — The MRI protocol will include standard anatomical, functional, and diffusion imaging, and spectroscopy sequences.
Behavioral: clinical assessments — Several clinical assessments will be performed to evaluate the recovery of motor functions. Initially and for screening, the cognitive ability will be assessed using the Montreal Cognitive Assessment (MoCA), and visuospatial neglect will be assessed using the Star Cancellation Test (SCT). eligible participants that meet all inclusion criteria will undergo a series of clinical function tests during each test session (t1-t4) to assess clinical outcomes.
  Groups: brain ischemic stroke patients

SUMMARY:
The investigator aims to find a correlation between brain structure and activity and spontaneous recovery of motor function following brain ischemic stroke by Analysis of MRI scans. The research includes stroke patients and healthy patients (control group).

DETAILED DESCRIPTION:
The recovery process, especially the recovery of motor functions after an ischemic stroke, differs from one person to another. In recent years, there is more evidence of spontaneous biological recovery (SBR), which is independent of training or rehabilitation-induced recovery, throughout the post-stroke subacute phase. However, the neural basis associated with motor function in this recovery phase remains unknown. We believe that the research results may help to explain the neural mechanism which promotes or inhibits recovery.

ELIGIBILITY:
Inclusion Criteria:

1. age between 21 years old and 80 years old
2. admission to the hospital 2-14 days after a first ischemic stroke, confirmed by CT, MRI or neurological report
3. residual unilateral upper extremity weakness
4. ability to give informed consent and understand the tasks involved.

Exclusion Criteria:

1. younger than 21 years old or older than 80 years old
2. cognitive impairment, as seen by a score of <20/30 on the Montreal Cognitive Assessment (MoCA)
3. history of a physical or neurological condition that interferes with study procedures or assessment of motor function (e.g. severe arthritis, severe neuropathy, Parkinson's disease)
4. contraindication to transcranial magnetic stimulation (TMS), such as deep brain stimulators or skull defect, presence of other metal devices or objects in the head, or a pacemaker
5. inability to sit in a chair and perform upper limb exercises for one hour at a time
6. inability to lie down in the MRI scanner for an hour
7. participation in another upper extremity rehabilitative therapy study during the study period
8. terminal illness
9. social and/or personal circumstances that interfere with the ability to return for therapy sessions and follow-up assessments
10. pregnancy
11. severe visuospatial neglect, as seen by a score of <44/54 on the Star Cancellation Test.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thirty stroke patients (experimental group) will be recruited from Sheba Medical Center, and 30 healthy age and gender-matched participants (control group) with no history of neurological impairments will be recruited from the community for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Neurochemical concentration levels as revealed by MRS scans. Including GABA, Glu and GSH. | Baseline GABA/ GLU/ GSH at <=2 weeks from stroke event (t1), change from Baseline GABA/ GLU/ GSH at 4 weeks (t2), change from Baseline GABA/ GLU/ GSH at 8 weeks (t3), change from Baseline GABA/ GLU/ GSH at 12 weeks (t4)
Clinical measures- Arm Research Action Test (ARAT) | Baseline ARAT at <=2 weeks from stroke event (t1), change from Baseline ARAT at 4 weeks (t2), change from Baseline ARAT at 8 weeks (t3), change from Baseline ARAT at 12 weeks (t4)
  The patient is seated at a table and is asked to perform tasks involving handling physical objects, on the table, with different properties (size, weight, shape, etc.).
Clinical measures- Fugl-Meyer Upper Extremity (FM-UE) | Baseline FM_UE at <=2 weeks from stroke event (t1), change from Baseline FM_UE at 4 weeks (t2), change from Baseline FM_UE at 8 weeks (t3), change from Baseline FM_UE at 12 weeks (t4)
  FM-UE- Administrator instructs patient to perform a series of physical tasks, also involves passive eliciting of reflexes for assessment.

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | Baseline MAS at <=2 weeks from stroke event (t1), change from Baseline MAS at 4 weeks (t2), change from Baseline MAS at 8 weeks (t3), change from Baseline MAS at 12 weeks (t4)
  Relevant limbs are passively manipulated through various degrees of range of motion while making observations of muscle tone.
Semmes-Weinstein Monofilament Examination (SWME) | Baseline SWME at <=2 weeks from stroke event (t1), change from Baseline SWME at 4 weeks (t2), change from Baseline SWME at 8 weeks (t3), change from Baseline SWME at 12 weeks (t4)
  Nylon filaments of different diameters are applied perpendicularly to the palmar surface of the index finger until the filament bends. The threshold is determined by the smallest diameter that is perceived.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No